CLINICAL TRIAL: NCT03322774
Title: Sleep To Reduce Incident Depression Effectively
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Big Health Inc. (Industry); University of Michigan (Other)
Responsible Party: Principal Investigator, Christopher Drake, Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: IRB 11586
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Insomnia, Primary; Major Depressive Disorder; Rumination
Keywords: Stepped Care
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major; Rumination Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Attention Control (Sham Comparator): This group receives sleep hygiene education, which serves as a credible control intervention to digital cognitive behavioral therapy for insomnia (dCBT-I). This intervention mimics the web-based patient contact inherent in dCBT-I but is inert with respect to sleep outcomes.
  Interventions: Behavioral: Sleep Hygiene Education Control
- Stepped Care Model (Experimental): This group receives digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) through the third party program, "Sleepio." Following initial treatment with dCBT-I, individuals who do not experience remission of their insomnia will begin treatment with face-to-face Cognitive Behavioral Therapy for Insomnia with a trained staff member in behavioral sleep medicine.
  Interventions: Behavioral: digital Cognitive Behavioral Therapy for Insomnia; Behavioral: face-to-face Cognitive Behavioral Therapy for Insomnia
- Stepped Care Model Control (Sham Comparator): This group receives digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) through the third party program, "Sleepio." Following initial treatment with dCBT-I, individuals who do not experience remission of their insomnia will receive sleep hygiene education, serving as a credible control intervention for comparison to the Stepped Care Model.
  Interventions: Behavioral: digital Cognitive Behavioral Therapy for Insomnia; Behavioral: Sleep Hygiene Education Control
- digital CBT-I (Experimental): This group receives digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) through the third party program, "Sleepio." Treatment includes weekly sessions of CBT-I administered over the internet in hour-long video sessions. Daily sleep diaries are recorded online for individual tailoring of treatment.
  Interventions: Behavioral: digital Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: digital Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia administered online through the "Sleepio" program. Treatment utilizes sleep restriction, stimulus control, and cognitive therapy. Treatment is administered through 6 weekly, hour-long online video sessions with an animated figure called "The Prof," which delivers the treatment.
  Other Names: Sleepio; dCBT-I
  Arms: Stepped Care Model; Stepped Care Model Control; digital CBT-I
Behavioral: face-to-face Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia administered by experienced staff trained in behavioral sleep medicine. Treatment utilizes sleep restriction, stimulus control, and cognitive therapy. Treatment is administered through 6 weekly, hour-long face-to-face sessions with an experienced staff member trained in behavioral sleep medicine.
  Other Names: CBT-I
  Arms: Stepped Care Model
Behavioral: Sleep Hygiene Education Control — Participants are provided with information about good sleep hygiene through 6 weekly emails. Participants practice good sleep hygiene as part of their sleep routine. In Step 1, sleep hygiene control will be exclusively online. In Step 2, sleep hygiene control includes an in-person, face-to-face component.
  Arms: Attention Control; Stepped Care Model Control

SUMMARY:
This project will assess the effectiveness of a stepped-care model (i.e. digital Cognitive Behavioral Therapy for Insomnia (dCBT-I) followed by face-to-face CBT-I) in improving severity of insomnia and sleep outcomes in an insomnia cohort. This project will also investigate the effectiveness of this stepped-care model in prevention of major depressive disorder, and will test rumination as a mediator of treatment response.

DETAILED DESCRIPTION:
This project will assess the acute and long-term effectiveness of dCBT-I on Research Domain Criteria (RDoC) sleep parameters: Insomnia Severity Index (ISI), sleep onset latency, and wake after sleep onset in an insomnia cohort including those at elevated risk for depression (e.g. low SES, minority). This will be tested by administering internet-based dCBT-I to people with insomnia and adding face-to-face CBT-I in non-remitters, as well as comparing the RDoC sleep outcomes to an attention control group post-treatment and at 1- and 2-year follow-ups. This study will also determine the acute and long-term effectiveness of face-to-face CBT-I in non-responders to dCBT-I on RDoC sleep outcomes relative to a comparison group post-treatment and at 1- and 2-year follow-ups.

This study will also determine the effects of dCBT-I and CBT-I using a stepped-care model for prevention of major depressive disorder incidence and relapse across 2 years. Specifically, rate of depression of both dCBT-I and CBT-I will be compared to a control group.

This study will also evaluate changes in rumination as a modifiable behavior (post-treatment) that mediates the effect of insomnia treatment on depression risk.

ELIGIBILITY:
Inclusion Criteria:

* Determination of Insomnia (ISI > 14)
* And no clinically significant depressive symptoms (Quick Inventory of Depressive Symptomatology < 11)

Exclusion Criteria:

* Age < 18
* Current use of antidepressants for depression
* Bipolar or Seizure disorders
* Known sleep disorders other than insomnia (e.g. obstructive sleep apnea, narcolepsy, restless leg syndrome).
* Current DSM-5 major depressive disorder at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1237 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Preventing major depressive disorder development with dCBT-I/CBT-I stepped care treatment for insomnia. | 1 and 2 years after initial randomization.
  Clinical interview by phone administered by trained personnel to determine DSM-5 major depressive disorder incidence and relapse. Major depressive disorder will specifically be determined by the structured clinical interview for DSM-5 (SCID-5) at 1- and 2-year follow-ups. Antidepressant history in the past 1 year is collected via online-administered surveys at 1- and 2-year follow-ups.
Effectiveness of Stepped Care model of dCBT-I/CBT-I for insomnia remission. | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Insomnia remission rates based on the Insomnia Severity Index. Total score range 0-28 with higher scores meaning more insomnia. Remission = ISI < 8.
Mediation of Depression Prevention by Reducing Rumination (Nocturnal rumination) | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Rumination as measured by the Pre-Sleep Arousal Scale, Cognitive factor. Scores range from 8 to 40 with higher scores indicating more rumination. Treatment-related changes in rumination will be operationalized as changes from pre- to posttreatment.

SECONDARY OUTCOMES:
Mediation of Depression Prevention by Reducing Rumination (Depressive rumination) | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Rumination as determined by the Rumination Response Scale. Scores range from 22-88 with higher scores indicating higher depressive rumination. Treatment-related changes in rumination will be operationalized as changes from pre- to posttreatment.
Mediation of Depression Prevention by Reducing Rumination (Worry) | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Rumination as determined by the Penn State Worry Questionnaire. Scores range from 16-80 with higher scores indicating greater worry. Treatment-related changes in rumination will be operationalized as changes from pre- to posttreatment.
Mediation of Depression Prevention by Reducing Rumination (Transdiagnostic) | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Rumination as determined by the Perseverative Thinking Questionnaire. Scores range from 15-75 with higher scores indicating greater perseverative thinking. Treatment-related changes in rumination will be operationalized as changes from pre- to posttreatment.
Reducing subclinical depressive symptoms with dCBT-I/CBT-I stepped care treatment for insomnia. | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Depressive symptoms as measured by the Quick Inventory of Depressive Sympatomatology, 16 item self report version. Reductions in depressive symptoms will be operationalized as (1) pre to posttreatment changes, (2) pretreatment to 1-year follow-up changes, and (3) pretreatment to 2-year follow-up changes.
Socioeconomic status as a moderator of depression prevention after stepped care insomnia treatment. | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Low socioeconomic status will be defined as annual household income < $20,000. Stepped care treatment will be less effective for preventing depression for patients in poverty as compared to patients above the the poverty line.
Racial minority identification as a moderator of depression prevention after stepped care insomnia treatment. | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Race will be self reported by patients. Stepped care treatment will be less effective for preventing depression for patients who self-identify as racial minorities (e.g., non-Hispanic black) relative to non-Hispanic white patients.
Stepped care insomnia treatment of dCBT-I and CBT-I will significantly improve sleep parameters. | Baseline, upon treatment completion, and then 1 and 2 years after initial randomization.
  Sleep parameters as captured by self-reported sleep onset latency, wake after sleep onset, and sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Drake, PhD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Medical Center - Columbus, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drake CL, Kalmbach DA, Cheng P, Ahmedani BK, Peterson EL, Joseph CLM, Roth T, Kidwell KM, Sagong C. Sleep to Reduce Incident Depression Effectively (STRIDE): study protocol for a randomized controlled trial comparing stepped-care cognitive-behavioral therapy for insomnia versus sleep education control to prevent major depression. Trials. 2022 Dec 1;23(1):967. doi: 10.1186/s13063-022-06850-4. PMID 36457045

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03322774/Prot_SAP_002.pdf